CLINICAL TRIAL: NCT02518347
Title: Effects of Freeze-dried Strawberries on Systemic Markers of Inflammation and Knee Function in Participants With Osteoarthritis (OA)
Brief Title: Strawberries and Knee Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, Oklahoma State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HE1517
Record Dates: First submitted 2015-07-30; First posted 2015-08-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDS-Strawberry (Experimental): Freeze-dried strawberry powder (50g/d)
  Interventions: Dietary Supplement: FDS-Strawberry
- Placebo (Placebo Comparator): Powder matched for carbohydrates and fiber in the strawberries
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: FDS-Strawberry — Natural frozen and dried strawberries
  Arms: FDS-Strawberry
Dietary Supplement: Placebo — Placebo powder matched for carbohydrates and fiber in the strawberries
  Arms: Placebo

SUMMARY:
The proposed study aims to examine the hypothesis that strawberry supplementation will lower serum biomarkers of inflammation and improve knee function in patients with symptomatic osteoarthritis (OA).

DETAILED DESCRIPTION:
The investigators propose the following two specific aims in a randomized crossover placebo-controlled trial in participants with two or more features of the metabolic syndrome and symptomatic osteoarthritis in this 12-week efficacy study:

Aim 1: To assess the effects of strawberries on biomarkers of inflammation [serum levels of C-reactive protein: CRP; inflammatory cytokines: interleukin-6: IL-6; interleukin 1β: IL-1β; tumor necrosis factor-alpha: TNFα] Aim 2: To assess the effects of strawberries on knee function as assessed by overall musculoskeletal examination and pain score (ICOAP, KOOS and HAQ-DI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee osteoarthritis
* Must have waist circumference >35 inches for women and >40 inches for men

Exclusion Criteria:

* Cancer
* Heart disease
* Smoking
* Berry allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | six months
Inflammatory Biomarkers in Serum | six months

CONTACTS AND LOCATIONS:
Overall Officials: ARPITA BASU, PHD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States